CLINICAL TRIAL: NCT07095777
Title: Study on the Recovery of Visual Perceptual Function Dysfunction in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Lixia Feng, Chief physician, Doctoral supervisor, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJ2022-09-48
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Retinopathy (DR); Visual Perception
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual perceptual learning group (Experimental)
  Interventions: Procedure: visual perceptual learning
- control group (No Intervention)

INTERVENTIONS:
Procedure: visual perceptual learning — Participants in the VPL group performed 40 minutes of daily monocular training at home for three months, with follow-up evaluations conducted at 1 month and 3 months after training initiation.
  Arms: visual perceptual learning group

SUMMARY:
Investigators aim to investigate the effectiveness of visual perceptual learning on visual perceptual function in participants with diabetic retinopathy and to provide novel therapeutic insights for visual functional rehabilitation in diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe non-proliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy(PDR) prior to treatment(17)
* prior pan retinal laser photocoagulation (PRP) at least 4 weeks before enrollment or vitreoretinal surgery at least 8 weeks before enrollment
* stable clinical condition
* best-corrected visual acuity (BCVA) > 1.0 logMAR (equivalent to a Snellen visual acuity of < 20/200)
* clear refractive media
* age ≤ 65 years
* ability to comprehend the examination and training procedures

Exclusion Criteria:

* significant refractive media opacity
* psychiatric disorders, chronic alcoholism and traumatic brain injury
* new-onset vitreous hemorrhage, myopia, strabismus, amblyopia, glaucoma and macular diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
contrast sensitivity | From enrollment to the end of treatment at 12 weeks
  The contrast sensitivity measurements include grating acuity, first-order motion stimulus perception sensitivity, second-order stationary stimulus perception sensitivity and second-order motion stimulus perception sensitivity, which represent the reciprocal of the contrast threshold.

SECONDARY OUTCOMES:
The Low Vision Quality of Life Questionnaire | From enrollment to the end of treatment at 12 weeks
  This instrument has demonstrated high reliability and validity, and is sensitive to changes in visual function among individuals with vision loss. The minimum value is 25 and the maximum value is 125. Higher scores indicate better quality of life.

OTHER OUTCOMES:
The Hospital Anxiety and Depression Scale | From enrollment to the end of treatment at 12 weeks
  The scale aims to measure anxiety and depression levels in hospital patients with high reliability and validity. The Hospital Anxiety and Depression Scale (HADS) provides separate scores for anxiety (HADS-A) and depression (HADS-D), each ranging from 0 to 21. A lower score indicates a lesser degree of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations. Participants did not consent to data sharing in the informed consent form.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT07095777/Prot_SAP_000.pdf